CLINICAL TRIAL: NCT06432868
Title: Effects of Solarplast (R) Supplementation on Biomarkers of Muscle Damage, Inflammation and Recovery of Physical Performance Following High-intensity Resistance Exercise
Brief Title: Solarplast (R) Supplementation Effects Following High-intensity Resistance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Adam Jajtner, Associate Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 927
Record Dates: First submitted 2024-04-29; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solarplast (R) (Active Comparator): 100mg/day of Solarplast (R) supplementation (28 days).
  Interventions: Dietary Supplement: Solarplast (R)
- Placebo (Placebo Comparator): 100mg/day of Placebo (maltodextrin (98.8%) and medium chain triglycerides (1.2%)).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Solarplast (R) — Daily supplementation for 28 days prior to heavy resistance exercise.
  Arms: Solarplast (R)
Dietary Supplement: Placebo — Daily supplementation for 28 days prior to heavy resistance exercise.
  Arms: Placebo

SUMMARY:
The primary goal of this investigation is to assess whether Solarplast (R) supplementation will improve recovery following heavy resistance exercise in active adults. The primary questions to be addressed are:

Does Solarplast (R) decrease muscle damage and inflammation associated with heavy resistance exercise?

Does Solarplast (R) reduce the decline in performance associate with heavy resistance exercise?

Researchers will compare Solarplast (R) to a placebo (a look-alike substance that contains no active ingredients) to see if Solarplast (R) is effective at improving recovery.

Participants will be asked to:

Take Solarplast (R) or placebo daily for 4 weeks

Visit the laboratory at least once per week to receive their supplement

Report to the lab for 3 consecutive visits following supplementation to complete a heavy resistance training session and follow-up testing.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally-active (participated in at least 2 weight training workouts per week over the previous year) and participates in at least 3h of total structured exercise/week as determined by the health and activity questionnaire.
* Subject is judged by the Investigator to be healthy and free of any physical limitations (determined by health and activity questionnaire)
* Subject has a body mass index of 18.0-34.9 kg/m2, inclusive
* Subject is willing to maintain habitual diet throughout the study period
* Subject is willing to abstain from dietary supplementation throughout the duration of the study.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators

Exclusion Criteria:

* Subject is currently or will be enrolled in another clinical trial.
* Subject is a habitual consumer of tea/antioxidants defined as > 8 oz/day of either green or black tea within the 14 days prior to the screening visit.
* Subject has a history or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder.
* Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Subject is unable to perform physical exercise (determined by health and activity questionnaire)
* Subject is engaged in an extreme diet including but not limited to, Atkins, South Beach, Intermittent Fasting, etc.
* Subject is allergic to the study product or placebo
* Subject is taking any other nutritional supplement or performance enhancing drug (determined from health and activity questionnaire)
* Subject has any chronic illness that causes continuous medical care
* Taking any type of prescription or over-the-counter medication including but not limited to corticosteroids, non-steroidal anti-inflammatory drugs, and antibiotics within the 14 days prior to the screening visit.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Creatine Kinase Activity | Acute changes following exercise for 48 hours
  Marker of Muscle Damage

SECONDARY OUTCOMES:
Myoglobin Concentration | Acute changes following exercise for 24 hours
  Marker of Muscle Damage
Vertical Jump Height | Acute changes following exercise for 48 hours
  Measure of Performance Change
Mean Squat Velocity | Acute changes following exercise for 48 hours
  Measure of Performance Change
Peak Isometric Muscle Force | Acute changes following exercise for 48 hours
  Measure of Performance Change
Rate of Force Development | Acute changes following exercise for 48 hours
  Measure of Performance Change
Ratings of Perceived Soreness | Acute changes following exercise for 48 hours
  Visual Analog Scale (1-100mm; low values indicate reduced soreness)
Ratings of Perceived Fatigue | Acute changes following exercise for 48 hours
  Visual Analog Scale (1-100mm; low values indicated reduced fatigue)

OTHER OUTCOMES:
Rate of Muscular Fatigue | Acute changes following exercise for 48 hours
  Measure of Performance Change
Rate of Muscular Fatigue | Change in Resting Values over 4 weeks of supplementation
  Measure of Performance Change
Lactate Dehydrogenase Activity | Acute changes following exercise for 48 hours
  Marker of Muscle Damage
Cortisol Concentration | Acute changes following exercise for 48 hours
  Circulating Marker of Stress
Cortisol Concentration | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Stress
Glutathione (GSH) Activity | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Oxidative Stress
Glutathione (GSH) Activity | Acute changes following exercise for 48 hours
  Circulating Marker of Oxidative Stress
Total Antioxidant Capacity | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Oxidative Stress
Total Antioxidant Capacity | Acute changes following exercise for 48 hours
  Circulating Marker of Oxidative Stress
Interleukin 6 (IL-6) Concentration | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Inflammation
Interleukin 6 (IL-6) Concentration | Acute changes following exercise for 48 hours
  Circulating Marker of Inflammation
Interleukin 10 (IL-10) Concentration | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Inflammation
Interleukin 10 (IL-10) Concentration | Acute changes following exercise for 48 hours
  Circulating Marker of Inflammation
Tumor Necrosis Factor - alpha (TNFa) Concentration | Change in Resting Values over 4 weeks of supplementation
  Circulating Marker of Inflammation
Tumor Necrosis Factor - alpha (TNFa) Concentration | Acute changes following exercise for 48 hours
  Circulating Marker of Inflammation
Rate of Force Development | Change in Resting Values over 4 weeks of supplementation
  Measure of Performance Change
Peak Muscle Force | Acute changes following exercise for 48 hours
  Measure of Performance Change
Vertical Jump Height | Change in Resting Values over 4 weeks of supplementation
  Measure of Performance Change

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University - Exercise Science & Exercise Physiology, Kent, Ohio, United States